CLINICAL TRIAL: NCT04421924
Title: Optimizing Periinterventional Coagulation Management of Patients Undergoing a Transjugular Intrahepatic Portosystemic Shunt Implantation: A Prospective Randomized Cohort Study
Brief Title: Periinterventional Coagulation Management of Patients Undergoing a TIPS
Acronym: TIPSprosp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TIPS-prospective
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombelastogram (TEG) (Experimental): Patients in the TEG group will receive prothrombin complex concentrates (PCC) at a dose of 10 IE/kg of ideal body weight, when R-time was greater than 40 minutes (2400 sec) and they will receive platelet transfusion in the amount of 1 apheresis unit when MA was below 30 mm.
  Interventions: Procedure: thrombelastogram
- Standard of Care (SOC) (Experimental): In the SOC group, patients will receive PCC at the dose of 10 IE /kg of ideal body weight when the PT is below 50% and/or INR>1.8 and/or received platelet transfusion in the amount of 1 apheresis when platelet count is below 50 G/L
  Interventions: Procedure: standard of care

INTERVENTIONS:
Procedure: thrombelastogram — Patients in the TEG group will receive prothrombin complex concentrates (PCC) at a dose of 10 IE/kg of ideal body weight, when R-time was greater than 40 minutes (2400 sec) and they will receive platelet transfusion in the amount of 1 apheresis unit when MA was below 30 mm
  Arms: Thrombelastogram (TEG)
Procedure: standard of care — 2) In the SOC group, patients will receive PCC at the dose of 10 IE /kg of ideal body weight when the PT is below 50% and/or INR>1.8 and/or received platelet transfusion in the amount of 1 apheresis when platelet count is below 50 G/L
  Arms: Standard of Care (SOC)

SUMMARY:
Assess whether a pre-interventional thrombelastography guided algorithm for assessing and correction of coagulation status in cirrhotic patients is safe and effective

DETAILED DESCRIPTION:
Transjugular intrahepatic portosystemic shunt (TIPS) is a very effective procedure to treat complications of portal hypertension in liver cirrhosis. TIPS implantation is indicated in cirrhotic patients to treat or prevent portal hypertensive bleeding and to treat refractory ascites.

During this procedure an artificial connection between portal vein and hepatic vein is placed via an image-guided endovascular approach. Although the procedure is very effective and reasonably safe, several complications can occur.

Due to the underlying cirrhosis, morbidity and mortality of TIPS is high, with a 30-day mortality between 7 and 20%. Procedural site complications (transhepatic and transvenous access), bleeding, development of hepatic encephalopathy or other organ complications and stent complications comprise a considerable risk to the patients, however, the improvement of mortality, renal function and liver function outweighs the risks of the procedure. Optimal patient selection and preoperative preparation is crucial to avoid complications of this procedure.

In liver cirrhosis, coagulation disturbances are common. In hepatic insufficiency, a balanced reduction in the levels of most of pro- and anticoagulant proteins produced in the liver does not impair thrombin generation until levels are quite low. However, the ability of the coagulation system to tolerate or recover from an insult is markedly impaired in liver disease. This allows the coagulation system to be more easily tipped into a state favouring either haemorrhage or thrombosis. The American Gastroenterology Association has recently published best practice advices to manage coagulation in cirrhosis. This review concludes that commonly used global coagulation tests are not optimal to assess the risk of bleeding in cirrhosis. A randomized controlled trial showed, that the use of thrombelastography (TEG) to assess coagulation in cirrhosis resulted in a significantly lower usage of blood products with no increase in bleeding rates.

The bleeding risk for TIPS implantation is not well studied, ranging from 0.6-4.3% of fatal bleeding complications in older uncontrolled case series. No evidenced-based recommendations exist for the correction of coagulation abnormalities before TIPS - and the few existing recommendations are not backed with evidence but rather "eminence based". Currently, global tests of coagulation (prothrombin time and platelet count) are used to guide coagulation correction. Mostly, cut-offs without sufficient evidence (PT >50%/ INR >1.8 and platelets >50 G/L) are used for correction of coagulation.

Also, the risk of stent thrombosis needs to be considered, therefore "blind" substitution of clotting factors or platelet transfusions is not advisable. Unfortunately, the study by De Pietri et al. (6) did only include one patient undergoing TIPS (in the standard of care (SOC) arm), therefore it is yet unknown, whether TEG is useful for guiding the correction of coagulation abnormalities in cirrhosis.

The aim of this trial is to assess, whether TEG guided pre-interventional assessment and correction of coagulation in cirrhotic patients is safe and effective

The study will be performed as a single-center, open-label, randomized prospective cohort study

ELIGIBILITY:
inclusion criteria

* Liver cirrhosis
* >18 years
* Indication for TIPS implantation
* Ability to sign informed consent exclusion criteria
* Contraindications against TIPS implantation
* Hepatocellular carcinoma BCLC D
* Ongoing bleeding
* pre-existing anticoagulant therapy at time of inclusion
* administration of blood products within 1 week prior to the enrolment
* Other malignancies that lead to an impaired 90-day survival
* Inherit blood clotting disorders
* Hepatic encephalopathy grade 3 or 4
* any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
blood product requirement | 2 days
  Amount of blood products (coagulation factors and platelet transfusions) transfused for pre-interventional correction of coagulation status

SECONDARY OUTCOMES:
Bleeding | 90 days
  Rate of bleeding complications (BARC criteria)
complications | 90 days
  Rate of transfusion related complications
Mortality | 90 days
  Mortality rate
Modified TIPS Score (MOTS) | 90 days
  Predictive power of modified TIPS score (MOTS) using the routine parameter, bilirubin, urea and INR; values range from 0-3, high score means worse outcome
Factor XIII | 2 days
  Comparison of measured FXIII activity levels with TEG parameters (alpha-angle, K-time, MA) for assessing feasibility of TEG in predicting deficiency of FXIII activity in these specific group of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No